CLINICAL TRIAL: NCT03201783
Title: A Randomized Trial Comparing the Effect of Immediate Versus Delayed Frozen-thawed Embryo Transfer Following a Stimulated IVF Cycle
Brief Title: Immediate Versus Delayed FET Following a Stimulated IVF Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShangHaiIVG
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2019-09

CONDITIONS: Fertilization in Vitro; Embryo Transfer
Keywords: frozen-thawed embryo transfer; time interval

STUDY DESIGN:
Masking Description: No masking because of the nature of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate group (Other): the intervention: immediate frozen-thawed embryo transfer (FET) which means FET will be performed in the first cycle following the stimulated IVF cycle
  Interventions: Other: immediate frozen-thawed embryo transfer
- delayed group (Other): the intervention: delayed frozen-thawed embryo transfer (FET) which means FET will be performed at least in the second cycle following the stimulated IVF cycle
  Interventions: Other: delayed frozen-thawed embryo transfer

INTERVENTIONS:
Other: immediate frozen-thawed embryo transfer — Frozen-thawed embryo transfer will be performed in the first cycle following the stimulated IVF cycle
  Arms: immediate group
Other: delayed frozen-thawed embryo transfer — Frozen-thawed embryo transfer will be performed at least in the second cycle following the stimulated IVF cycle
  Arms: delayed group

SUMMARY:
Information regarding the optimal timing for frozen-thawed embryo transfer (FET) following a stimulated in vitro fertilization (IVF) is lacking. One option is to perform FET in the first cycle following the stimulated IVF cycle, i.e. immediate transfer. Another option is to postpone FET for at least one menstrual cycle, i.e. delayed transfer. This randomized study aims to compare the ongoing pregnancy rate of immediate versus delayed FET following a stimulated IVF cycle.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≤43 years at the time of IVF/ICSI treatment Undergoing IVF with a standard stimulation At least one frozen embryo or blastocyst The first FET cycle following ovarian stimulation in IVF/ICSI

Exclusion Criteria:

* Use of mild stimulation or natural cycle for IVF/ICSI treatment Severe ovarian hyperstimulation syndrome during IVF/ICSI treatment Preimplantation genetic diagnosis treatment Use of donor oocytes Presence of hydrosalpinx which is not surgically treated or endometrial polyp on scanning during ovarian stimulation

Ages: 20 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 724 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
ongoing pregnancy | viable pregnancy beyond gestation 12 weeks
  viable pregnancy beyond gestation 12 weeks

SECONDARY OUTCOMES:
Positive hCG level | A blood pregnancy test is performed 14 days after the FET
  the result of serum β-hCG ≥10 mIU/mL.
clinical pregnancy | presence of intrauterine gestational sac on ultrasound at 6 weeks of pregnancy
  presence of intrauterine gestational sac on ultrasound
biochemical pregnancy: | positive blood pregnancy test not followed by clinical pregnancy during 12 weeks gestation
  positive blood pregnancy test not followed by clinical pregnancy
implantation rate | number of gestational sacs per embryo transferred during 4 weeks of pregnancy
  number of gestational sacs per embryo transferred
multiple pregnancy | multiple pregnancy beyond gestation 12 weeks
  more than one intrauterine sacs on scanning
ectopic pregnancy | ectopic pregnancy during 12 weeks gestation
  pregnancy outside the uterine cavity
miscarriage | the loss of a pregnancy before 22 weeks gestation
  the loss of a pregnancy before 22 weeks gestation
live birth rate | a live birth after 22 weeks gestation
  the rate of live births per cycle
birth weight | a live birth after 22 weeks gestation
  birth weight of the baby delivered

CONTACTS AND LOCATIONS:
Overall Officials: XIAOXI SUN, PHD, Principal Investigator — Shanghai JiAi Genetics & IVF Institute
Locations (1):
- ShangHai JIAI Genetics&IVF Institute, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification (text, tables, figures, and appendices) and study protocol will be shared. Data will be available when beginning 3 months and ending 5 years following article publication. To achieve aims in the approved proposal, researchers who provide a methodologically sound proposal will be shared with.Data will be made available by the following way. Proposals should be directed to lihe198900@163.com. And data are available for 5 years at a third party website (link to be included after the article publication).

REFERENCES:
- [Background] Santos-Ribeiro S, Siffain J, Polyzos NP, van de Vijver A, van Landuyt L, Stoop D, Tournaye H, Blockeel C. To delay or not to delay a frozen embryo transfer after a failed fresh embryo transfer attempt? Fertil Steril. 2016 May;105(5):1202-1207.e1. doi: 10.1016/j.fertnstert.2015.12.140. Epub 2016 Jan 21. PMID 26806686
- [Background] Santos-Ribeiro S, Polyzos NP, Lan VT, Siffain J, Mackens S, Van Landuyt L, Tournaye H, Blockeel C. The effect of an immediate frozen embryo transfer following a freeze-all protocol: a retrospective analysis from two centres. Hum Reprod. 2016 Nov;31(11):2541-2548. doi: 10.1093/humrep/dew194. Epub 2016 Sep 8. PMID 27609984
- [Background] Lattes K, Checa MA, Vassena R, Brassesco M, Vernaeve V. There is no evidence that the time from egg retrieval to embryo transfer affects live birth rates in a freeze-all strategy. Hum Reprod. 2017 Feb;32(2):368-374. doi: 10.1093/humrep/dew306. Epub 2016 Dec 16. PMID 27986819
- [Background] Volodarsky-Perel A, Eldar-Geva T, Holzer HE, Schonberger O, Reichman O, Gal M. Cryopreserved embryo transfer: adjacent or non-adjacent to failed fresh long GnRH-agonist protocol IVF cycle. Reprod Biomed Online. 2017 Mar;34(3):267-273. doi: 10.1016/j.rbmo.2016.11.013. Epub 2016 Dec 16. PMID 28041829
- [Derived] Li H, Sun X, Yang J, Li L, Zhang W, Lu X, Chen J, Chen H, Yu M, Fu W, Peng X, Chen J, Ng EHY. Immediate versus delayed frozen embryo transfer in patients following a stimulated IVF cycle: a randomised controlled trial. Hum Reprod. 2021 Jun 18;36(7):1832-1840. doi: 10.1093/humrep/deab071. PMID 33885131
- [Derived] Li H, Li L, Lu X, Sun X, Ng EHY. Comparison of the effect of immediate versus delayed transfer following a stimulated IVF cycle on the ongoing pregnancy rate of frozen-thawed embryo transfer cycles: a study protocol for a randomised controlled trial. BMJ Open. 2018 May 17;8(5):e020507. doi: 10.1136/bmjopen-2017-020507. PMID 29773699